CLINICAL TRIAL: NCT01202604
Title: Prospective, Observational Study for the Maintenance Treatment of Patients With Bipolar Disorder I and II in Greece.
Brief Title: A Study Evaluating the Efficacy of Administered Maintenance Treatments in Bipolar Disorder I and II.
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NGR-DUM-2010/1
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder I and II; mood event; manic or depressive; Greece
MeSH Terms: conditions — Bipolar Disorder; Mania

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Outpatients with bipolar disorder I or II (as per DSM-IV): The percentage of patients who experience a relapse episode during the first 9 months after a mood event (manic or depressive).

SUMMARY:
The primary objective of the study is to evaluate the efficacy of administered maintenance treatments in bipolar disorder I and II, defined as the percentage of patients who experience a relapse episode during the first 9 months after a mood event (manic or depressive).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who experienced the last acute mood episode during the last 2 months and are in euthymic state (YMRS score ≤12 and HAM-D score ≤12) for at least two weeks
* Diagnosis of bipolar disorder I or II (as per DSM-IV), with or without rapid cycling
* Subjects who have been treated with at least one atypical antipsychotic for the management of an acute mood event (manic or depressive) as monotherapy or in combination with other medication
* Provision of informed consent prior to study participation

Exclusion Criteria:

* Subjects fulfilling criteria for diagnosis of any other psychiatric condition (except from bipolar disorder I or II), as per DSM-IV Axis Ι, concomitant organic mental disorder or mental retardation
* Subjects who have received treatment with a depot
* Substance abuse or dependence (with the exception of nicotine dependence), as defined by DSM-IV criteria
* Inability of subjects to comply with the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients diagnosed with bipolar disorder I or II (as per DSM-IV), who have received therapy with at least one atypical antipsychotic for the acute episode and whose treating physician has considered they have entered the maintenance phase.
Sampling Method: Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The proportion of patients (n, %) who will experience a relapse episode (manic, hypomanic, depressive, mixed) | During the first 9 months after the acute mood episode or in case of relapse occurrence.

SECONDARY OUTCOMES:
Description of administered treatments for the management of the acute phase of bipolar disorder [mood stabilizers (n,%), antidepressants (n,%), and antipsychotics (n,%)]. | 4 months and 9 months after the acute mood episode or in case of relapse occurrence
Description of management of relapse episodes in patients previously receiving treatment during the maintenance phase | In all visits - during the whole study period (9 months)
YMRS total score, HAM-D total score | At baseline and final visit (9 months after the acute mood episode)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Panagiotis Pontikis, Study Director — AstraZeneca S.A. Greece
Locations (33):
- Greece (33):
  - Research Site, Aigio, Achaias
  - Research Site, Ag. Paraskevi, Attikis
  - Research Site, Athens, Attikis
  - Research Site, Chaïdári, Attikis
  - Research Site, Drapetsona, Attikis
  - Research Site, Elefsina, Attikis
  - Research Site, Glyfada, Attikis
  - Research Site, Ilissia, Attikis
  - Research Site, Kifissia, Attikis
  - Research Site, Koropí, Attikis
  - Research Site, Marousi, Attikis
  - Research Site, N. Kosmos, Attikis
  - Research Site, Pangrati, Attikis
  - Research Site, Petroúpolis, Attikis
  - Research Site, Piraeus, Attikis
  - Research Site, Thebes, Attikis
  - Research Site, Vironas, Attikis
  - Research Site, Ag. Nikolaos, Crete
  - Research Site, Agrinio, Etoloakarnania
  - Research Site, Arta, Etoloakarnania
  - Research Site, Alexandroupoli, Evros
  - Research Site, Lamia, Fhiotidos
  - Research Site, Amaliáda, Ilias
  - Research Site, Karditsa, Karditsas
  - Research Site, Katerini, Katerinis
  - Research Site, Kavala, Kavalas
  - Research Site, Sparti, Lakonias
  - Research Site, Edessa, Pellas
  - Research Site, Giannitsá, Pellas
  - Research Site, Preveza, Prevezis
  - Research Site, Serres, Serres
  - Research Site, Thessaloniki, Thessalonikis
  - Research Site, Trikala, Trikalon